CLINICAL TRIAL: NCT01127919
Title: Training Interventions and Genetics of Exercise Response (TIGER)
Acronym: TIGER
Status: Completed | Type: Observational
Sponsor: Molly S. Bray (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Molly S. Bray, Professor of Public Health, University of Texas at Austin
Organization: University of Texas at Austin (Other)
Other Study IDs: R01DK062148 (NIH); R01DK062148 (NIH)
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Exercise Response
Keywords: Exercise; Activity; Adherence; Genetics
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood components and DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Low Commitment: Group 1 participants will take a 1-credit hour course that involves exercise training only.
  Interventions: Behavioral: Aerobic Exercise Training
- High Commitment: Group 2 participants will take a 3-credit hour course that involves exercise training plus an online cognitive component that provides information on fitness and health topics and includes quizzes and other written course work
  Interventions: Behavioral: Aerobic Exercise Training; Other: Cognitive Component
- Non-Exercise: Group 3 participants will take the cognitive component of the formal course but will not partake in the formalized exercise program for a period of 35 weeks.
  Interventions: Other: Cognitive Component

INTERVENTIONS:
Behavioral: Aerobic Exercise Training — 40 minutes, 3 times a week for 35 weeks.
  Groups: High Commitment; Low Commitment
Other: Cognitive Component — Provide general information about health and fitness
  Groups: High Commitment; Non-Exercise

SUMMARY:
Obesity established in adolescence strongly predicts obesity for the remainder of adult life, and the consequences are potentially devastating, characterized by a lifelong burden of co-morbid conditions and depression. This study will provide an exposure to physical activity that is designed to teach and empower sedentary college age individuals to become physically active. The investigators will evaluate whether such exposure can result in lasting changes in exercise behavior and body composition. The study will also provide a better understanding of the genetic factors that influence persistence in an exercise program and that influence whole body response to exercise training. Altering the course of obesity in adolescence has the potential to reduce the adult prevalence of obesity and consequently attenuate the public health burden of overweight and obesity in the investigators population.

DETAILED DESCRIPTION:
Among the greatest public health concerns today is the rapid rise in obesity in the pediatric population, which now exceeds 18% in children (6-11 y) and 17% in adolescents (12-19 y), while obesity among young adults (20-39 y) approaches 30%. Though much has been learned regarding the regulation of body weight and the development of adiposity, the prevalence of obesity continues to rise, demonstrating that even today the factors that predict healthy weight maintenance remain poorly understood. In fact, the transition from overweight adolescent to obese adult is almost inevitable, with the probability of obesity in adulthood exceeding 50% among children >13 years of age whose BMI percentiles meet or exceed the 95th percentile for age and gender. But what if we could deter the expected transition from overweight adolescent to obese adult and intervene on a young person at a critical time when he/she is beginning to feel empowered by independence? This is the essence of the Training Interventions and Genetics of Exercise Response (TIGER) Study. The TIGER Study began in 2003 with the goal of identifying genetic factors that influence physiologic response to exercise training, while introducing sedentary college age individuals to regular exercise. Subjects in the TIGER Study currently underwent 30 weeks (2 semesters) of exercise training, 3 days per week for 40 minutes at 65-85% of age-predicted maximum heart rate. More than 80% of subjects lost weight or maintained their weight within 2 kg, and only 18% of subjects gained more than 2 kg. We have identified preliminary associations between gene variation and exercise dropout in the first phase of the study, and in phase 2 of the TIGER study, we will build on these observations. We will focus on three primary areas of investigation: 1) formal evaluation of the TIGER Study intervention protocol to achieve long-term change in the participants; 2) investigation of gene expression patterns in skeletal muscle and subcutaneous adipose tissue as a strategy for identifying genes related to exercise response; and 3) investigation of the association between genetic variation and exercise adherence. Subjects will undergo 35 weeks of exercise training based on the established TIGER protocol, and subjects will be re-contacted 6, 12, and 24 months following completion of the study protocol and questioned regarding current exercise habits and body weight. In addition, genetic analysis of candidate genes related to exercise behavior and neural signaling will be undertaken in order to identify genetic factors that may influence exercise adherence. Finally, patterns of gene expression in subcutaneous adipose, skeletal muscle, and peripheral leukocytes will be analyzed at baseline and following exercise training in order to identify factors that influence physiologic change consequent to exercise training. Results from this study are designed to enlighten our current understanding of how and why individuals respond and/or persist in exercise, with the ultimate goal of formulating better and more efficacious interventions for obesity.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years old
* Healthy
* sedentary at baseline

Exclusion Criteria:

* any medical or physical contra-indication for exercise (as indicated by the subject's physician) and/or
* any known metabolic or endocrine disorder associated with alterations in body composition (e.g., lipodystrophy).
* Refusal to consent for the use of their DNA for genetic research.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The target for phase 2 of the TIGER study is a student, age 18-30, who has not engaged in moderate physical activity more than 30 minutes per week for the previous 30 days and who is not actively limiting his/her caloric intake by dieting. It is planned to enroll a total of 3,200 subjects from student populations at the University of Houston (UH) and the University of Alabama at Birmingham (UAB) and representative of the race/ethnicity distribution of the respective campuses. Approximately 2,400 subjects will participate in the exercise protocol (600/yr for four years). A control group (200/yr for four years) will also be recruited that will not participate in the formal exercise for at least 35 weeks, but will be given the option of completing the formal exercise program after that time.
Sampling Method: Non-Probability Sample
Enrollment: 3773 (Actual)
Dates: Start 2010-07; Primary Completion 2016-05 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Exercise Response | 15 Weeks
  Physiologic variables measured pre and post exercise intervention
Gene Expression | 15 Weeks
  Changes in the expression of genes following exercise training
Adherence | 15 Weeks
  Retention versus drop-out from the exercise protocol
Genotyping | 15 Weeks
  Characterization of candidate genes related to exercise response

CONTACTS AND LOCATIONS:
Overall Officials: Molly Bray, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Houston, Houston, Texas